CLINICAL TRIAL: NCT01290471
Title: Phase 1, Open Label Study to Assess the Safety and Tolerability of U3 1565 in Subjects With Advanced Solid Malignant Tumors
Brief Title: Study to Assess the Safety and Tolerability of U3-1565 in Subjects With Advanced Solid Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U31565-A-U101
Record Dates: First submitted 2011-02-02; First posted 2011-02-07 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Advanced Solid Malignant Tumors; Advanced Ovarian Cancer
MeSH Terms: interventions — U3-1565

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 Dose Escalation (Experimental): Dose escalation of U3 1565 will follow a modified 3+3 study design with a starting intravenous (IV) dose of 2 mg/kg. A maximum of 2 new subjects will receive their first dose of U3-1565 per 24-hour period during the dose-escalation phase. Subsequent escalating doses of 8, 16, and 24 mg/kg are planned. Three to 6 subjects will be enrolled in 4 sequential dose level cohorts.
  Interventions: Drug: U3-1565
- Part 2a Dose Expansion (Experimental): For Part 2a, 6 or 12 subjects with advanced solid malignant tumors will be enrolled and treated at the MTD or MAD to further define the safety and tolerability of U3-1565. These additional subjects are expected to permit the detection of relatively rare toxicities that would not likely be observed during the dose escalation part of the study, whose 3+3 design implies a maximum of 6 subjects only will be treated at the MTD or MAD. Six subjects will be treated; however, if toxicities meeting the definition of DLT are observed during the first cycle of treatment, 6 more subjects will be treated for a total of 12 subjects.
  Interventions: Drug: U3-1565
- Part 2b Dose Expansion and Anti-tumor Impact (Experimental): For Part 2b, up to 30 subjects with advanced solid malignant tumors, with a preference for those with advanced ovarian cancer, will be enrolled and treated at the MTD or MAD. This number of subjects should allow demonstrating U3-1565 has anti-tumor impact by showing treatment-induced changes in pharmacodynamic biomarkers and clinical activity. Ovarian cancer may be more likely to be impacted by U3 1565 than other tumors, considering that in this cancer, high levels of HB-EGF have been associated with an unfavorable clinical outcome. Six subjects will be initially treated; at which point, a safety analysis will be conducted after these initial subjects have completed the first cycle of treatment, to allow the reevaluation of the appropriateness of the dosing level.
  Interventions: Drug: U3-1565

INTERVENTIONS:
Drug: U3-1565 — U3 1565 will be provided as a sterile, frozen solution. Each glass vial will contain 1.1 mL (1 mL extractable) of study medication with a concentration of 100 mg/mL. U3 1565 will be diluted in a final volume of 100 mL and administered by continuous IV infusion over 60 minutes. Infusion times can be extended to a maximum of 120 minutes for subjects unable to tolerate the 60 minute infusion.

SUMMARY:
This is a Phase 1, open label study to assess the safety and tolerability of U3 1565, determine maximum tolerated dose (MTD) or establish maximum administered dose (MAD) safety and tolerability.

DETAILED DESCRIPTION:
This study will be conducted in 2 phases: a dose-escalation phase corresponding to Part 1 and a dose-expansion phase articulated in 2 concomitant parts (i.e., Parts 2a and 2b).

All parts of this study are single arm and open label. In all parts, tumor assessments will be performed at screening and every 3 cycles thereafter, while the subject remains on study. U3-1565 clinical activity will be assessed measuring tumor response by physical examination and imaging according to RECIST version 1.1, if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented advanced solid malignant tumor refractory to standard treatment or for which no standard treatment is available.
* Evaluable tumor for all parts of the study and, only for enrollment in Part 2b, measurable tumor per RECIST version 1.1. However, subjects with advanced ovarian cancer may be enrolled in Part 2b even if they do not have a tumor measurable per RECIST version 1.1, as long as they have circulating levels of CA125 higher than 35 U/mL.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1.
* Men or women >= 18 years of age.
* Willing to provide pre-existing diagnostic or resected tumor samples, such as paraffin embedded sections, if available.
* Willing, only for enrollment in Part 2b, to provide tumor biopsies before and after treatment.
* For female subjects, is postmenopausal (no menstrual period for a minimum of 12 months) or surgically sterile or, if otherwise of childbearing potential, has a negative urine or serum pregnancy test at entry into the study, uses maximally effective birth control during the course of the study, and is willing to use contraception for 6 months following the last study drug administration.
* For male subjects, is surgically sterile or willing to use a double barrier contraception method upon enrollment, during the course of the study, and for 6 months following the last study drug administration.
* Able to comprehend, sign, and date current Institutional Review Board- (IRB) approved informed consent form (ICF - including Health Insurance Portability and Accountability Act [HIPAA] authorization, if applicable) before performance of any study-specific procedures or tests.

Exclusion Criteria:

* History of lymphoma, leukemia, or other hematopoietic malignancy.
* History of human immunodeficiency virus (HIV) positivity. HIV testing is not required for establishing eligibility.
* History of bleeding diathesis.
* History of idiosyncratic reactions to antibody drug products.
* History of stem cell or bone marrow transplant.
* History of myocardial infarction (MI) within 6 months before enrollment, symptomatic congestive heart failure (CHF; New York Heart Association > Class II), unstable angina or unstable cardiac arrhythmia requiring medication
* History of clinically significant pulmonary disease after receiving epidermal growth factor receptor- (EGFR) targeting agents.
* Any concomitant medical condition that would increase the risk of toxicity, in the opinion of the Investigator or Sponsor.
* Clinically active brain metastases defined as symptomatic or requiring treatment with steroids or anti-convulsants.
* Unresolved toxicities from prior anti-cancer therapy defined as toxicities, except alopecia, not yet resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 Grade =< 1 or baseline values. Subjects with chronic Grade 2 toxicities may be eligible at the discretion of the Investigator or Sponsor (eg, Grade 2 chemotherapy-induced neuropathy).
* Mean QTcF (Fridericia's correction) intervals > 450 msec for male subjects and > 470 msec for female subjects, based on screening electrocardiogram (ECG).
* Moderate to severe cardiac valvular abnormalities identified by echocardiography at screening.
* Hematological values, as follows:

Absolute neutrophil count (ANC) < 1.5 X 109/L Platelet count < 100 X 109/L Hemoglobin (Hb) < 9 g/dL - Renal function, as follows: Creatinine > 1.5 X upper limit of normal (ULN) or creatinine clearance < 60 mL/min, as calculated using the modified Cockcroft Gault equation.

- Hepatic function, as follows: Aspartate aminotransferase (AST) > 3 X ULN (if liver metastases are present, > 5 X ULN).

Alanine aminotransferase (ALT) > 3 X ULN (if liver metastases are present, >= 5 X ULN)

* Bilirubin > 1.5 X ULN
* Coagulation function, as follows:

Prothrombin time (PT) or partial thromboplastin time (PTT) > 1.5 X ULN

* Anti-cancer therapy, including antibody, retinoid, or hormonal treatment, within 3 weeks before enrollment. Prior and concurrent use of hormone replacement therapy, use of gonadotropin-releasing hormone modulators for prostate cancer, and use of somatostatin analogs for neuroendocrine tumors are permitted.
* Therapeutic radiation treatment within 4 weeks or palliative radiation treatment within 2 weeks before enrollment, as long as radiation toxicities have resolved to NCI CTCAE grade =< 1 or baseline values.
* Major surgery within 4 weeks before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number (percent) of subjects experiencing adverse events (AEs) after treatment with U3-1565 | 6 months
  Number (percent) of subjects experiencing adverse events (AEs) after treatment with U3-1565

SECONDARY OUTCOMES:
determine the maximum tolerated dose (MTD) or tolerability of maximum administered dose (MAD). | 12 months
Greatest percent reduction in the sum of longest diameters (SLD) of measurable tumors, if applicable, after U3 1565 treatment | 24 months
Changes in pharmacodynamic biomarkers in blood and other body fluid specimens | 24 months
  Changes in pharmacodynamic biomarkers in blood and other body fluid specimens (such as soluble HB-EGF and CA125 in serum and ascites) and tumor biopsies after U3 1565 treatment.
Changes in tumor perfusion and vascularity after U3-1565 treatment using Dynamic Contrast Enhanced Magnetic Resonance Imaging (DCE MRI) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Senaldi, MD, PhD, Study Director — Daiichi Sankyo
Locations (4):
- United States (4):
  - Karmanos Cancer Center, Detroit, Michigan
  - Univ. Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee